CLINICAL TRIAL: NCT04181684
Title: Pilot Study of Laser Interstitial Thermal Therapy Followed By Hypofractionated Radiation Therapy for Treatment of Recurrent Gliomas.
Brief Title: LITT Followed by Hypofractionated RT for Recurrent Gliomas
Acronym: GCCC 19140
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Keep Punching Foundation (Unknown)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00088569
Record Dates: First submitted 2019-11-24; First posted 2019-11-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Brain Tumor; Glioma; Neoplasms
Keywords: Gliomas, Laser Interstitial Thermal Therapy, Brain, Brain Tumor, Radiotherapy, Proton Therapy, Hypofractionated Radiation Therapy, Malignant, Glioblastoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental: LITT with Hypofractionated radiation therapy (Experimental): Laser interstitial thermal therapy (LITT) followed by hypo-fractionated radiation therapy, 35Gy/10 fractions.
  Interventions: Device: Procedure: LITT; Radiation: Hypo-Fractionated Radiation Therapy

INTERVENTIONS:
Device: Procedure: LITT — This procedure is done under MRI guidance and employs low-powered thermal energy to achieve tumor ablation through coagulation.
  Other Names: Laser Interstitial thermal therapy
Radiation: Hypo-Fractionated Radiation Therapy — Treatments will be delivered once daily on consecutive treatment days (typically 5 fractions per week). Radiation therapy simulation is to be performed within 10 days of the LITT procedure.

SUMMARY:
The purpose of this study is to evaluate the treatment regimen of using Laser Interstitial Thermal Therapy (LITT) and Hypo-fractionated Radiation Therapy to treat patients with recurrent gliomas.

DETAILED DESCRIPTION:
Radiation therapy is preferably used as an adjunct to surgery for patients with a newly diagnosed or recurrent glioblastoma. LITT offers an alternative to surgical resection, and due to its minimally invasive nature, does not delay initiating radiation therapy. Another advantage of LITT prior to radiation therapy is the ability to obtain a tissue diagnosis of recurrent tumor prior to initiating radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of a WHO Grade II-IV glioma with radiographic evidence of recurrent or progressive tumor

   * Patient must have received prior radiation therapy for initial treatment of glioma
   * Patients with any number of recurrences are allowed as long as the patient has not undergone re-irradiation
2. Brain MRI with contrast demonstrates an enhancing tumor ≤ 6 cm in largest diameter within 60 days prior to registration
3. History and physical including neurological exam within 30 days prior to registration
4. Karnofsky performance status ≥ 60% within 30 days prior to registration
5. Age ≥ 22 years old
6. Minimum interval since completion of prior radiation treatment is 8 weeks

   * Patients will only receive re-irradiation if pathology from LITT is consistent with recurrent tumor
7. Patients must have signed an approved informed consent
8. Patients with the potential for pregnancy or impregnating their partner must agree to practice effective contraceptive methods to avoid conception while on study and for 6 months after study completion.
9. Female patients of child-bearing potential must have a negative pregnancy test within 28 days prior to study registration.

Exclusion Criteria:

1. Patients that are not surgical candidates for stereotactic biopsy or laser ablation
2. Patients with impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * History or presence of serious uncontrolled ventricular or significant arrhythmias.
   * Any of the following within 6 months prior to registration: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cerebrovascular accident, transient ischemic attack , pulmonary embolism
3. Infratentorial tumor or evidence of leptomeningeal spread
4. Inability to undergo a MRI
5. Pregnant or breast-feeding women

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 2 years
  To complete protocol treatment without undue treatment-related acute toxicity in recurrent or progressive glioma subjects undergoing LITT followed by hypofractionated radiation therapy.

SECONDARY OUTCOMES:
Progression-free survival at 6 months | 2 Years
  To describe progression-free survival rate in subjects with recurrent or progressive gliomas treated with Laser Interstitial Thermal Therapy
Median progression-free survival | 2 Years
  To describe median progression-free survival rate in subjects with recurrent or progressive gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
Median overall survival | 2 years
  To describe median progression-free survival rate in subjects with recurrent or progressive gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
1-year overall survival | 2 years
  To describe 1 year overall survival rate in subjects with recurrent or progressive gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
Overall response rate | 2 years
  To describe overall response survival rate in subjects with recurrent or progressive gliomas treated with Laser Interstitial Thermal Therapy followed by hypofractionated radiation therapy.
Quality of Life before, during, and after treatment | 2 years
  Patient reported quality of life impact from undergoing LITT followed by hypofractionated radiation therapy using the M.D. Anderson Symptom Inventory- Brain Tumor (MDASI-BT) questionnaire.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - UCH Kaufman Cancer Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland

IPD SHARING:
Plan to Share IPD: No